CLINICAL TRIAL: NCT02314897
Title: Left Ventricular Pacing to Prevent Iatrogenic Tricuspid Regurgitation Caused by Conventional Right Ventricular Pacing: a Pilot Study
Brief Title: Left Ventricular Pacing to Prevent Iatrogenic TR Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/00258
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2017-04

CONDITIONS: Tricuspid Valve Insufficiency; Sick Sinus Syndrome
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LV pacing (Experimental): Left ventricular pacing lead implanted via coronary sinus
  Interventions: Device: LV pacing
- RV pacing (Active Comparator): Conventional right ventricular pacing lead.
  Interventions: Device: RV pacing

INTERVENTIONS:
Device: LV pacing — Left ventricular pacing lead implanted via the coronary sinus.
  Arms: LV pacing
Device: RV pacing — Conventional right ventricular pacing.
  Arms: RV pacing

SUMMARY:
Background and Aims Pacemaker implantation for treating bradyarrhythmias typically involves placing a pacing lead through the tricuspid valve (TV) into the right ventricular (RV) apex. It is now known that tricuspid regurgitation (TR) frequently results from this and may lead to increased morbidity or mortality. Recently, left ventricular (LV) pacing through an epicardial vein via the coronary sinus has been widely practiced due to the advent of biventricular pacing. This lead does not cross the TV, potentially reducing the risk of TV dysfunction and may also reduce the risk of LV dysfunction. The investigators hypothesize that LV pacing will prevent the onset of new TR or worsening of pre-existing TR in patients undergoing pacemaker implantation.

Methods Patients receiving a pacemaker for sick sinus syndrome (n=20) with an LV ejection fraction <40% will be randomly allocated to receive either conventional RV pacing or LV pacing via the coronary sinus. Serial 2D and 3D transthoracic echocardiography will be performed before implantation, one day post implantation, then at 1 week, 1 month, 6 months and 1 year. The primary endpoints will be new onset TR and the diagnosis of at least moderate TR. Other endpoints include biventricular function, ventricular dyssynchrony, complications of device implantation, mortality and major cardiovascular events.

DETAILED DESCRIPTION:
We hypothesize that left ventricular pacing via a coronary sinus approach can reduce the incidence of significant tricuspid regurgitation after pacemaker implantation in patients with normal left ventricular function.

The aim of this study is to compare the degree of tricuspid regurgitation caused by pacemaker implantation between the conventional techniques of implanting a ventricular lead implanted in the right ventricular apex versus implanting a ventricular lead in a left ventricular epicardial vein via a coronary sinus approach.

The secondary objective of our study is to evaluate whether left ventricular pacing is also less likely to cause ventricular dyssynchrony and dysfunction than right ventricular apical pacing.

This study is a single centre randomised clinical pilot study comparing 2 different lead implantation techniques to be assessed using both imaging techniques and follow up for clinical outcomes.

(i) Proposed study interventions The procedures in both arms of the study will be identical except for where the ventricular lead is placed. All parts of these procedures, including all the implanting equipment and pacing leads are standard routine clinical practice. The left ventricular leads used in this study are routinely used for pacing the left ventricle in patients receiving biventricular pacemakers or defibrillators for heart failure.

The implant site will be the left or right prepectoral region and venous access will be via either an axillary or subclavian vein approach. These choices will be left to the implanting physician's discretion. Once venous access has been established successfully the patient will then be randomly allocated to either of the study arms.

Patients randomized to have an LV lead will have a long coronary sinus sheath inserted which will be used to perform an occlusive venogram of the coronary sinus to determine if there are veins suitable for left ventricular lead placement. Those in the left ventricular pacing arm will instead have a left ventricular epicardial pacing lead placed as apically as possible in a large calibre left ventricular branch of the coronary sinus.

Patients in the right ventricular apical pacing arm will have an endocardial active fixation pacing leads placed in the right ventricular apex in the conventional manner.

Patients in both arms will then go on to have a right atrial active fixation lead placed in the right atrial appendage.

(ii) Methods for protecting against other sources of bias All patients referred to our Arrhythmia Service will be assessed for suitability to take part in this study. Once recruited, study subjects will be block randomised in a 1:1 fashion to either conventional right ventricular lead implantation or left ventricular coronary sinus lead implantation. They will be blinded to their allocation during the course of this study to remove any bias.

Assessment of the echocardiograms will be performed by 2 investigators who are not blinded to the patient's treatment allocation. This is because the pacemaker lead is nearly always well visualised during echocardiographic studies making blinding impossible. However, the main outcomes of this study will be quantitative measures of TR and biventricular function derived from 3D echocardiography rather than qualitative measures used in previous studies and this will protect against bias that may be caused by the echocardiogram assessors knowing the allocation of the patients. The studies will also be assessed for interobserver and intraobserver variability to look for the likelihood of bias.

(iii) Duration of follow up period Patients will be seen post discharge at 1 week for wound care and at 1 months, 6 months and 12 months for pacemaker checks in the pacemaker clinic.

(iv) Frequency and duration of follow-up The scheduled follow up is as follows. Note that all transthoracic echocardiography studies will include both 2D and 3D echocardiography

1. Pre implant: transthoracic echocardiography
2. Pacemaker implantation: randomisation when venous access is achieved. Blood samples taken for biomarker assays.
3. Post implant day 1: Pacemaker check, transthoracic echocardiography
4. Post implant week 1: Wound check, pacemaker check, transthoracic echocardiography
5. Post implant month 1: Wound check, pacemaker check, transthoracic echocardiography
6. Post implant month 6: Pacemaker check, transthoracic echocardiography, blood samples taken for biomarker assays.
7. Post implant month 12: Pacemaker check, transthoracic echocardiography

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing dual chamber permanent pacemaker implantation for sick sinus syndrome. This is defined as symptomatic sinus node dysfunction manifest as sinus pauses or excessive sinus bradycardia and is diagnosed on continuous ECG monitoring or ambulatory ECG recording (Holter study).
2. Aged ≥21 years and able to give informed consent. The age limit is so that all patients are able to give informed consent personally.

Exclusion Criteria:

1. Left ventricular ejection fraction <40%. 2. Mobitz Type 2 second degree atrioventricular block, 2:1 atrioventricular block, high degree atrioventricular block or complete heart block.

1. Life expectancy less than 1 year due to medical co-morbidities.
2. Previous mechanical prosthetic tricuspid valve replacement, precluding the implantation of a right ventricular apical lead.
3. Tricuspid regurgitation that is at least moderate in severity.
4. Complex congenital heart disease precluding the placement of either a right ventricular apical lead or left ventricular lead via the coronary sinus
5. Vascular or coronary sinus anatomy unfavourable to either conventional RV lead or left ventricular lead implantation as confirmed on a coronary sinus venography at the time of implantation.
6. Pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Development of moderate or worse TR post implantation | 6 months
  At least moderate of worsening of tricuspid regurgitation at 6 months post implantation on echocardiography

SECONDARY OUTCOMES:
Biventricular ventricular function and dyssynchrony | 6 months
  Echocardiographically determined LV function, RV function, interventricular and intra ventricular dyssynchrony at 6 months.
Major cardiovascular events | 6 months
  Cardiovascular mortality, hospitalizations, heart failure, stroke, MI
All cause mortality | 6 months
  All cause mortality
Biomarkers of heart failure | 6 months
  Change in plasma concentrations over 6 months of NT-proBNP, hsTnT and GDF15
Lead performance parameters | 6 months
  Change in lead parameters over 6 months, including sensed R wave amplitude, impedance, capture threshold.
Procedural complications and device related complications | 6 months
  Procedural complications and device related complications

CONTACTS AND LOCATIONS:
Overall Officials: Toon Wei Lim, MBBS, PhD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore